CLINICAL TRIAL: NCT07025798
Title: The Impact of Compound Probiotic Freeze-dried Powder on Enhancing Gastrointestinal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20250616
Record Dates: First submitted 2025-06-16; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Tract
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wec120B group (Experimental)
  Interventions: Dietary Supplement: Probiotic
- Wec300B group (Experimental)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic strips with different strain formulas, Specification: 2g/bag. Storage method: Keep away from light, seal tightly, and store in a cool, dry place.

SUMMARY:
The primary objective of this study is to evaluate the effects of the compound probiotic freeze-dried powder on gastrointestinal function and its impact on gut microbiota, immune factors, inflammatory markers, and intestinal barrier function.

ELIGIBILITY:
Inclusion Criteria:

（1）Age: 18-65; （2）It conforms to the diagnostic criteria for gastrointestinal dysfunction formulated in the "Expert Consensus on Precision Health Communication in China - Guidelines for Citizens' Intestinal Health"; （3）Symptoms: Irregular defecation, loose or hard stools; Intestinal rumbling in the abdomen Abdominal distension Hiccups, belching; Severe intestinal flatulence; Abdominal pain Acid reflux and heartburn; Pain in the stomach or abdomen when hungry; Disgusting; (4) Signs: Abdominal pain and abdominal distension; Diarrhea and constipation Indigestion Gastric acid reflux Bad breath and farting smell; Skin problems The color and shape of the stool have changed.

-

Exclusion Criteria:

(1)Drugs that affect the intestinal flora (including antibacterial drugs, microecological preparations, intestinal mucosal protectants, traditional Chinese patent medicines, etc.) should be used continuously for more than one week within one month before screening; （2）Recent use of products with similar functions to the test product, which may interfere with the judgment of the study results; (3) use of antibiotics during illness; (3)Use of antibiotics during illness; (4)Resence of severe systemic diseases or malignant tumors; (5)allergy to any components of the probiotics used in the study; (6)women who are pregnant, breastfeeding, or planning to conceive in the near future.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Improvement of gastrointestinal symptoms | 4 weeks
  Bowel movement frequency improvement: use the "bowel movement frequency scale"

CONTACTS AND LOCATIONS:
Locations (1):
- School of Food and Bioengineering, Henan University of Science and Technology, Luoyang, Henan, China